CLINICAL TRIAL: NCT07170761
Title: Cross-sectional Biomarker Study for Vascular Calcification in Hemodialysis Patients
Brief Title: Biomarkers and Event Patterns of Vascular Disease in Hemodialysis
Acronym: HEMOcalc
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: LKH Feldkirch (Unknown); Elisabethinen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 34-322 ex 21/22
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Vascular Disease; CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder
MeSH Terms: conditions — Vascular Diseases; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parathyroid hormone (PTH) remains the central biomarker to classify CKD-metabolic bone disease (CKD-MBD) in hemodialysis patients. While PTH-values are known to be associated with adverse outcomes, interventional studies have failed to show a benefit of pharmacological modulation of PTH levels on hard clinical outcomes. To address this gap, the investigators explored alternative markers of bone metabolism, vascular calcification and inflammation in association to prospective event patterns.

ELIGIBILITY:
Inclusion Criteria:

* Stable hemodialysis > 3 months duration

Exclusion Criteria:

* Pregnancy
* Acute infections with antibiotic treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prevalent, chronic hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1, 2 and 3 years
  All-causes, the date of death will be recorded.

SECONDARY OUTCOMES:
Cause-specific mortality | 1, 2 and 3 years
  The cause of death will be recorded.
MACE | 1, 2 and 3 years
  The number of participants with, the date and cause of MACE (a composite outcome measure of non-fatal and fatal stroke, myocardial infarction, acute heartfailure and sudden cardiac death) will be recorded from medical record review.
The number of participants with hospitalisation for Infection | 1, 2 and 3 years
  The number and dates of hospitalisations for any infectious diseases (such as pneumonia, sepsis or urinary tract infection) will be recorded from medical record review.
The number of participants with hospitalisation for Heart failure | 1, 2 and 3 years
  The number and dates of hospitalisations for heart failure (such as acute heart failure or decompensated chronic heart failure) will be recorded from medical record review.
The number of participants with Fractures | 1, 2 and 3 years
  The number and dates of fractures (classified by anatomical site, such as hip, vertebral, or upper limb) will be recorded from medical record review.
The number of participants with Bleeding events | 1, 2 and 3 years
  The number and dates of bleeding events (classified as major or minor according to ISTH definition) will be recorded from medical record review.
The number of participants with Interventions for vascular diseases | 1, 2 and 3 years
  The number and dates of surgical and endovascular interventions (such as revascularization, bypass or amputation) for atherosclerotic cardiovascular diseases (such as coronary and peripheral artery disease) will be recorded from medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Eller, Univ.-Prof., Principal Investigator — Division of Nephrology, Department of Internal Medicine, Medical University of Graz, Graz, Austria
Locations (1):
- Medical University Graz, Graz, Styria, Austria